CLINICAL TRIAL: NCT01384851
Title: Therapeutic Efficacy of the Chronic Application of Tear Formulations for Dry Eye and Normal Subjects Under Conditions of Environmental Stress
Brief Title: Efficacy of the Chronic Application of Tear Formulations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Glasgow Caledonian University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Alan Tomlinson, Glasgow Caledonian University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AG9965-004
Record Dates: First submitted 2011-06-23; First posted 2011-06-29 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Next Generation Emulsion (Experimental): Next Generation Emulsion Multi-Dose Eye Drop (9963X) is a sterile, buffered, aqueous and emulsion topical ophthalmic product formulated for the relief of ocular surface irritation and symptoms of dryness. The Next Generation Emulsion 9963X formulation is an oil-in-water aqueous emulsion intended to replenish deficient aqueous and lipid components and stabilising the tear film.
  Interventions: Drug: Next Generation Emulsion
- Refresh Dry Eye Therapy (Active Comparator): A preserved multi-dose formulation for use in treating dry eye symptomatology. The key ingredients are Castor oil, Polysorbate 80, Carbomer 1342 and Glycerin. Refresh Dry Eye Therapy® Lubricant Eye Drops contains emulsified castor oil, which enhances the natural oily superficial tear layer on the ocular surface. By stabilizing and supplementing the lipid layer, castor oil may retard evaporation of surface moisture.
  Interventions: Drug: Refresh Dry Eye Therapy
- Refresh Contacts (Active Comparator): Solution contains carboxymethylcellulose sodium (carmellose), sodium chloride, boric acid, sodium borate, potassium chloride, calcium chloride, magnesium chloride, Purite®, sodium hydroxide, and purified water. This product is registered as a CE Mark medical device. Refresh Contacts Comfort drops providing soothing relief from tired, dry eyes. Although intended for contact lens wearers, the primary indication is for relief of dry eyes as is being studied in this investigation.
  Interventions: Drug: Refresh Contacts

INTERVENTIONS:
Drug: Next Generation Emulsion — One drop both eyes 4 times daily for two weeks
  Arms: Next Generation Emulsion
Drug: Refresh Dry Eye Therapy — One drop both eyes four times daily for two weeks
  Arms: Refresh Dry Eye Therapy
Drug: Refresh Contacts — One drop both eyes four times daily for two weeks
  Arms: Refresh Contacts

SUMMARY:
The purpose of this study is to determine the therapeutic effect of the chronic application of eye-drops on tear evaporation rate in dry eye and normal subjects exposed to a condition of environmental stress. The effect will be studied in terms of changes in tear physiology and the inflammatory biomarkers on the ocular surface.

DETAILED DESCRIPTION:
Environmentally induced dry eye is a condition which occurs in otherwise asymptomatic individuals in certain situations, for example with the use of computers, in overheated or air conditioned workplaces and in conditions of low humidity. The most common ocular complaints associated with these environments are burning, dryness, stinging, and grittiness. Although the exact cause of these symptoms is unknown, it is thought that increased tear evaporation rate due to low humidity plays a vital role. The changes in tear film physiology, which occurs in these environments, have traditionally been dealt with by the use of eye drops (particularly the highly viscous variety), which have been shown to be an effective therapeutic option in the treatment of environmental dry eye disease. Previous studies of the use of eye-drops of various formulations has shown improvements in tear physiology in mild to moderate dry eye patients with their use in both acute and chronic application protocols. In this study, an attempt was made to relate the effects on tear physiology induced by variations in environmental conditions to the beneficial effect produced by the use of eye-drops.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 79 years of age.
* Must understand and be able, willing and likely to fully comply with study procedures and restrictions.

Exclusion Criteria:

* Active ocular allergy
* Current contact lens wear
* Any topical ophthalmic drops within 1 week of initial screening visit.
* Started or changed the dose of chronic systemic medication known to affect tear production including, but not limited to antihistamines, antidepressants, diuretics, corticosteroids or immunomodulators within 30 days of initial screening visit.
* Systemic disease known to affect tear production or loss including, but not limited to thyroid eye disease, that has been diagnosed or has not been stable within 30 days initial of screening visit.
* Known hypersensitivity to any of the agents used in testing.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Tear Film Evaporation | Each subject will be followed for the duration of the study, an expected average of 8-9 weeks
  Tear film evaporation will be determined with a 'Servo-Med EP-Evaporimeter'. This measures the relative humidity and temperature at two sensors separated by a known distance, above the evaporative surface. The ocular surface evaporation will be calculated from measurements of fluid loss with the eyes open and closed while the subject sits with the eye covered by a modified goggle.

SECONDARY OUTCOMES:
Interferometry | Each subject will be followed for the duration of the study, an expected average of 8-9 weeks
  The structure and quality of the tear film will be assessed by observing the interference fringes of the lipid layer. Interferometry facilitated with a miniature slow motion video will be used. The grading system developed previously in our laboratory will be utilised to grade the tear film distribution. This grading system classifies the tear film structure on the basis of the distribution of tears after a blink. Measurements are made while the subject sits quietly and looks into the lens of the device.
Tear Film Osmolarity | Each subject will be followed for the duration of the study, an expected average of 8-9 weeks
  Tear film osmolarity was measured using an 'OcuSense TearLab Osmometer'. This employs a single use, disposable test card mounted to a collection pen, to obtain a small sample of tear fluid by passive capillary action from the inferior-temporal tear meniscus. The measurement of the electrical impedance is carried out within the pen. The pen is then docked into the reader, which calculates and displays the osmolarity result.
Non-invasive tear break up time | Each subject will be followed for the duration of the study, an expected average of 8-9 weeks
  The 'HIR-CAL Grid' system based on a modified Bausch and Lomb keratometer will be used. The 'HIR-CAL Grid'will be focused on the pre-corneal tear film and the time before first distortion of the grid image will be recorded. This will indicate the non-invasive tear break up time. Three measurements will be taken while the subject is instructed to blink and then to hold the eye open while the examiner watches the reflection from the tear film, and the mean calculated.
Tear sampling and bio-marker analysis | Each subject will be followed for the duration of the study, an expected average of 8-9 weeks
  Approximately 1 μl of tears will be collected from the subject's eye using a sterile micropipette.
  It will then be diluted in cytokine assay buffer and simultaneously analysed for biomarkers of ocular surface disease (cytokines) using the Luminex Beadlyte assay system. The bio-markers to be studied are included in the Human high sensitivity cytokine/chemokine kit (Millipore). These markers are associated with pro-inflammatory activation and have been previously studied in dry eye and other inflammatory conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tomlinson, DSc PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom